CLINICAL TRIAL: NCT06797674
Title: A Clinical Study to Evaluate the Effect of Multiple Doses of Efavirenz on Single-Dose Pharmacokinetics of MK-7602 in Healthy Participants
Brief Title: A Study of the Effect Efavirenz on the Plasma Levels of MK-7602 in Healthy Participants (MK-7602-005)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 7602-005
Record Dates: First submitted 2025-01-21; First posted 2025-01-28 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Healthy
MeSH Terms: interventions — efavirenz

STUDY DESIGN:
Intervention Model Description: Part 1 has a single arm. Part 2 will enroll participants in a crossover design, randomized between 6 different treatment sequences.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1: MK-7602 + Efavirenz (Experimental): Participants will be administered MK-7602 and efavirenz.
  Interventions: Drug: MK-7602; Drug: Efavirenz
- Part 2, Sequence 1: Fasted→Moderate-Fat Meal→Low-Fat Meal (Experimental): Participants will be administered MK-7602 in the fasted state, then with a moderate-fat meal, then with a low-fat meal.
  Interventions: Drug: MK-7602
- Part 2, Sequence 2: Fasted→Low-Fat Meal→Moderate-Fat Meal (Experimental): Participants will be administered MK-7602 in the fasted state, then with a low-fat meal, then with a moderate-fat meal.
  Interventions: Drug: MK-7602
- Part 2, Sequence 3: Moderate-Fat Meal→Low-Fat Meal→Fasted (Experimental): Participants will be administered MK-7602 with a moderate-fat meal, then with a low-fat meal, then in the fasted state.
  Interventions: Drug: MK-7602
- Part 2, Sequence 4: Moderate-Fat Meal→Fasted→Low-Fat Meal (Experimental): Participants will be administered MK-7602 with a moderate-fat meal, then in the fasted state, then with a low-fat meal.
  Interventions: Drug: MK-7602
- Part 2, Sequence 5: Low-Fat Meal→Fasted→Moderate-Fat Meal (Experimental): Participants will be administered MK-7602 with a low-fat meal, then in the fasted state, then with a moderate-fat meal.
  Interventions: Drug: MK-7602
- Part 2, Sequence 6: Low-Fat Meal→Moderate-Fat Meal→Fasted (Experimental): Participants will be administered MK-7602 with a low-fat meal, then with a moderate-fat meal, then in the fasted state.
  Interventions: Drug: MK-7602

INTERVENTIONS:
Drug: MK-7602 — Capsule
Drug: Efavirenz — Tablet
  Other Names: MK-0831
  Arms: Part 1: MK-7602 + Efavirenz

SUMMARY:
The goal of the study is to learn what happens to levels of MK-7602 in a healthy person's body over time. Researchers will compare what happens to MK-7602 in the body when it is given with or without another medicine called efavirenz, and when it is given with or without a meal.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Has a body-mass index (BMI) of 18 to 32 kg/m^2.

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* Has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and seizures) abnormalities or diseases.
* Has a history of cancer (malignancy)
* Has positive test(s) for hepatitis B surface antigen, hepatitis C antibodies, or human immunodeficiency virus (HIV)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of MK-7602 | At designated time points (up to 4 weeks)
  Blood samples will be collected to determine the AUC0-inf of MK-7602.
Area Under the Concentration-Time Curve from Time 0 to 24 hours (AUC0-24hrs) of MK-7602 | At designated time points (up to 4 weeks)
  Blood samples will be collected to determine the AUC0-24hr of MK-7602.
Maximum Plasma Concentration (Cmax) of MK-7602 | At designated time points (up to 4 weeks)
  Blood samples will be collected to determine the Cmax of MK-7602.
Time to Maximum Plasma Concentration (Tmax) of MK-7602 | Predose and at designated time points (up to 4 weeks)
  Blood samples will be collected to determine the Tmax of MK-7602.
Plasma Concentration at 24 Hours (C24) of MK-7602 | At designated time points (up to 4 weeks)
  Blood samples will be collected to determine the C24 of MK-7602.
Apparent Terminal Half-life (t1/2) of MK-7602 | At designated time points (up to 4 weeks)
  Blood samples will be collected to determine the t1/2 of MK-7602.

SECONDARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 10 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 10 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be reported.
Part 2: AUC0-Inf of MK-7602 | At designated time points (up to 4 weeks)
  Blood samples will be collected to determine the AUC0-inf of MK-7602.
Part 2: AUC0-24hrs of MK-7602 | At designated time points (up to 4 weeks)
  Blood samples will be collected to determine the AUC0-24hr of MK-7602.
Part 2: Cmax of MK-7602 | At designated time points (up to 4 weeks)
  Blood samples will be collected to determine the Cmax of MK-7602.
Part 2: Tmax of MK-7602 | Predose and at designated time points (up to 4 weeks)
  Blood samples will be collected to determine the Tmax of MK-7602.
Part 2: C24 of MK-7602 | At designated time points (up to 4 weeks)
  Blood samples will be collected to determine the C24 of MK-7602.
Part 2: t1/2 of MK-7602 | At designated time points (up to 4 weeks)
  Blood samples will be collected to determine the t1/2 of MK-7602.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Fortrea Clinical Research Unit Inc ( Site 0001), Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com